CLINICAL TRIAL: NCT00004420
Title: Study of Gammalinolenic Acid for Juvenile Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13314; UMASS-H-2703; UMASS-FDR001067
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-01

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: arthritis & connective tissue diseases; juvenile rheumatoid arthritis; rare disease
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis; Connective Tissue Diseases; Rare Diseases | interventions — gamma-Linolenic Acid

INTERVENTIONS:
Drug: gamma-Linolenic acid

SUMMARY:
OBJECTIVES:

I. Determine the efficacy and safety of gammalinolenic acid in the treatment of childhood arthritis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, cross over study of 12 months duration. Patients are stratified by type of juvenile rheumatoid arthritis (systemic onset vs pauciarticular disease vs polyarticular disease).

Patients are randomized to receive either gammalinolenic acid (GLA) or placebo (safflower seed oil) orally. Parents are asked to maintain the child's usual diet over the course of study.

Patients are followed at 3, 6, 9, and 12 months during study and at 6 months thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Juvenile rheumatoid arthritis (systemic onset, pauciarticular disease, and polyarticular disease)
* Active synovitis

--Prior/Concurrent Therapy--

* No more than 2 concurrent nonsteroidal antiinflammatory drugs
* No more than 2 concurrent second line agents (e.g., D-penicillamine, oral or injectable gold, antimalarials, methotrexate, sulfasalazine)
* Must have started second line agent at least 3 months prior to study
* Must be on stable doses of all medications for at least 1 month prior to study
* Prior prednisone allowed if started at least 3 months prior to study

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 1994-09; Study Completion 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Zurier, Study Chair — University of Massachusetts, Worcester